CLINICAL TRIAL: NCT07261813
Title: Chronic Obstructive Pulmonary Disease, Quality of Life, COPD Assessment Test, Nepal, Dyspnea, Spirometry
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of medicine, Maharagjung medical campus (Other)
Responsible Party: Principal Investigator, Abhishek Kumar Shah, Principal Investigator, Institute of medicine, Maharagjung medical campus
Other Study IDs: 353 (6-11) E2 077/ 078
Record Dates: First submitted 2025-11-14; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of Quality of life in COPD patients — This study does not involve a clinical intervention. Instead, it focuses on evaluating Quality of life of COPD patient using the COPD Assessment Test (CAT). It is a validated, patient-completed questionnaire designed to assess the impact of Chronic Obstructive Pulmonary Disease (COPD) on a patient's health status. It consists of eight simple questions, each scored from 0 to 5, covering symptoms such as cough, sputum production, chest tightness, breathlessness, activity limitation, confidence leaving home, sleep quality, and energy levels. The total score ranges from 0 to 40, with higher scores indicating a greater impact of COPD on the patient's daily life. A score of 0-10 suggests a low impact, 11-20 a medium impact, 21-30 a high impact, and 31-40 a very high impact. The CAT is easy to administer, typically taking less than two minutes to complete, and provides clinicians with a standardized way to monitor disease progression and evaluate treatment effectiveness.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterized by airflow limitation that is not fully reversible. The study "Quality of life among people living with Chronic Obstructive Pulmonary Disease- visiting spirometry center of Tribhuvan University Teaching Hospital, Kathmandu Nepal" aims to assess the quality of life (QOL) of COPD patients and the factors affecting it.

A cross sectional study will be performed among the patients visiting Spirometry center of Tribhuvan University Teaching Hospital, Kathmandu Nepal using Convenience Sampling. Ethical approval will be obtained from Institutional Review Board (IRB) of TUTH and written/verbal consent for data collection will be obtained from Teaching hospital authority as well as the respondents. CAT questionnaire will be used to assess quality of life and the Medical Research Council questionnaire will be used to assess the severity of dyspnea. Data management and analysis will be conducted through Statistical Package for Social Sciences (SPSS) version 26.0.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* Referred to the spirometry center of Tribhuvan University Teaching Hospital
* Confirmed diagnosis of COPD based on GOLD criteria: post-bronchodilator FEV1/FVC < 0.7

Exclusion Criteria:

* Unable to perform acceptable spirometry maneuvers
* Presence of significant respiratory diseases that can confound COPD assessment (e.g., asthma, bronchiectasis, active tuberculosis)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study enrolled participants aged 20 years or older who were referred to the spirometry center of Tribhuvan University Teaching Hospital. The primary inclusion criterion was a confirmed diagnosis of COPD based on the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria, defined as a postbronchodilator ratio of forced expiratory volume in one second to forced vital capacity (FEV1/FVC) < 0.70.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life (HRQoL) Score (COPD Assessment Test - CAT) | 1 month
  The COPD Assessment Test (CAT) score ranges from 0 to 40, with 0 indicating no impact and 40 indicating the worst impact on quality of life. Higher scores represent worse outcomes.

IPD SHARING:
Plan to Share IPD: No
Since this is an observational study focused on evaluating the quality of life of COPD patients, Individual Participant Data (IPD) will not be shared as part of the study's results. However, the aggregated findings, such as overall satisfaction scores and analysis of demographic factors influencing consent understanding, will be presented in the final study report.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-11-29): https://cdn.clinicaltrials.gov/large-docs/13/NCT07261813/Prot_SAP_ICF_000.pdf